CLINICAL TRIAL: NCT07145619
Title: Effect of Bilateral Ultrasound-Guided Transversus Abdominis Plane Block on Quality of Recovery in Cesarean Delivery Patients Receiving Intrathecal Morphine: A Prospective Observational Cohort Study
Brief Title: Effect of Bilateral Ultrasound-Guided TAP Block on Quality of Recovery in Cesarean Delivery Patients Receiving Intrathecal Morphine
Acronym: QoR-TAP
Status: Recruiting | Type: Observational
Sponsor: MEHMET GÖKHAN TAFLAN (Other)
Responsible Party: Sponsor-Investigator, MEHMET GÖKHAN TAFLAN, Principal Investigator, Specialist in Anesthesiology, Samsun University
Organization: Samsun University (Other)
Other Study IDs: ITMTAPObsQoRMT2025; GOKAEK2024/18/8 (Other: Samsun University)
Record Dates: First submitted 2025-08-14; First posted 2025-08-28 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Pain Management; Obstetric Anesthesia; Recovery From Anesthesia
Keywords: Cesarean delivery; Spinal anesthesia; Intrathecal morphine; Transversus abdominis plane block; Postoperative pain; Obstetric anesthesia; Quality of recovery
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ITM: Patients undergoing elective cesarean delivery under spinal anesthesia with 100 µg intrathecal morphine (ITM) as part of standard care. No additional regional block will be performed. Postoperative analgesia will be maintained with intravenous patient-controlled analgesia (IV PCA) using morphine, along with multimodal analgesia.Approximately 75 participants will be enrolled in this group
  Interventions: Other: Spinal Anesthesia with Intrathecal Morphine Only
- ITM + TAP: Patients undergoing elective cesarean delivery under spinal anesthesia with 100 µg intrathecal morphine (ITM) as part of standard care, plus bilateral ultrasound-guided transversus abdominis plane (TAP) block performed at the end of surgery. Postoperative analgesia will be maintained with intravenous patient-controlled analgesia (IV PCA) using morphine, along with multimodal analgesia.Approximately 75 participants will be enrolled in this group
  Interventions: Other: Spinal Anesthesia with Intrathecal Morphine plus Bilateral TAP Block

INTERVENTIONS:
Other: Spinal Anesthesia with Intrathecal Morphine Only — Elective cesarean delivery performed under spinal anesthesia with the addition of 100 micrograms intrathecal morphine (ITM) as part of standard clinical care. No additional regional block is performed. Postoperative analgesia is maintained with intravenous patient-controlled analgesia (IV PCA) morphine and multimodal analgesia, including scheduled paracetamol and NSAIDs as per institutional protocol.
  Groups: ITM
Other: Spinal Anesthesia with Intrathecal Morphine plus Bilateral TAP Block — Elective cesarean delivery performed under spinal anesthesia with the addition of 100 micrograms intrathecal morphine (ITM) as part of standard clinical care, plus bilateral ultrasound-guided transversus abdominis plane (TAP) block performed at the end of surgery. The TAP block will be performed in-plane with a high-frequency linear probe, using 0.25% bupivacaine, 20 mL per side, injected between the internal oblique and transversus abdominis muscles. Postoperative analgesia will be maintained with intravenous patient-controlled analgesia (IV PCA) morphine and multimodal analgesia, including scheduled paracetamol and NSAIDs.
  Groups: ITM + TAP

SUMMARY:
This prospective, assessor-blinded observational cohort study will investigate the effect of adding bilateral ultrasound-guided transversus abdominis plane (TAP) block to standard intrathecal morphine (ITM) analgesia on the quality of recovery in women undergoing elective cesarean delivery under spinal anesthesia. All participants will receive ITM as part of routine spinal anesthesia. The TAP group will receive an additional bilateral ultrasound-guided TAP block at the end of surgery, while the control group will not receive any additional block. Both groups will receive standardized postoperative analgesia with intravenous patient-controlled analgesia (IV PCA). The primary outcome is the quality of recovery at 24 hours postoperatively, measured using the validated Obstetric Quality of Recovery-10 (ObsQoR-10) questionnaire. Secondary outcomes include Numerical Rating Scale (NRS) pain scores, time to first breastfeeding, time to mobilization, time to hospital discharge, and total opioid consumption in the first 24 hours after surgery. Outcome assessors will be blinded to group allocation. The study aims to determine whether TAP block enhances functional recovery, reduces pain, and decreases analgesic requirements when used alongside ITM in cesarean delivery patients.

DETAILED DESCRIPTION:
Effective postoperative analgesia is essential for optimizing maternal recovery after cesarean delivery, promoting early mobilization, and supporting breastfeeding initiation. Spinal anesthesia with intrathecal morphine (ITM) is commonly used due to its long-lasting analgesia; however, it may not provide complete abdominal wall analgesia and can be associated with opioid-related side effects. The transversus abdominis plane (TAP) block is an ultrasound-guided regional anesthesia technique that provides somatic analgesia to the anterior abdominal wall by targeting the anterior rami of the thoracolumbar spinal nerves (T6-L1). When combined with ITM, TAP block may further improve recovery quality, reduce opioid requirements, and facilitate earlier return to daily activities.

In this prospective, assessor-blinded observational cohort study, all eligible patients undergoing elective cesarean delivery under spinal anesthesia at our institution will receive ITM as part of standard practice. Participants will be managed in two groups based on postoperative analgesia:

* TAP Group: Bilateral ultrasound-guided TAP block performed at the end of surgery in addition to ITM.
* Control Group: ITM only, without additional regional block.

Both groups will receive standardized postoperative analgesia via intravenous patient-controlled analgesia (IV PCA). Data will be collected prospectively, and the outcome assessor responsible for postoperative evaluation will be blinded to group allocation.

Primary Outcome:

* Quality of recovery at 24 hours postoperatively, measured using the Obstetric Quality of Recovery-10 (ObsQoR-10) questionnaire.

Secondary Outcomes:

* Numerical Rating Scale (NRS) pain scores
* Time to first breastfeeding
* Time to first mobilization
* Time to hospital discharge
* Total opioid consumption within the first 24 hours

By analyzing these parameters, the study aims to clarify whether the addition of TAP block to ITM-based analgesia can enhance recovery quality, improve functional outcomes, reduce pain intensity, and decrease opioid consumption in cesarean delivery patients. Findings from this research could inform best practice guidelines for postoperative pain management in obstetric anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18-45 years
* Singleton pregnancy
* ASA physical status II-III
* Scheduled elective lower segment cesarean delivery under spinal anesthesia with intrathecal morphine (ITM) as standard care
* Able to understand study procedures, provide written informed consent, and reliably use IV PCA
* Able to complete ObsQoR-10-T assessments (with trained assistance if needed)

Exclusion Criteria:

* Contraindication to spinal anesthesia or TAP block (e.g., infection at injection site, coagulopathy, allergy to local anesthetics)
* Chronic opioid use or opioid/alfa-2 agonist intolerance
* Severe preeclampsia, HELLP syndrome, significant hepatic or renal impairment
* Urgent or emergent cesarean section (Category 1)
* Cognitive impairment or communication difficulty preventing accurate assessment
* Prior major abdominal surgery (other than previous cesarean delivery)
* Body mass index (BMI) > 40 kg/m²
* Major psychiatric illness (e.g., major depressive disorder, generalized anxiety disorder, psychosis) that may affect pain perception or quality of recovery

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women undergoing elective cesarean delivery under spinal anesthesia with intrathecal morphine at a tertiary university hospital. Two observational cohorts will be followed: one receiving only intrathecal morphine and the other receiving intrathecal morphine plus bilateral ultrasound-guided TAP block.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
Obstetric Quality of Recovery-10 (ObsQoR-10) Score at 24 Hours Postoperatively | 24 hours after surgery
  Total score on the validated Turkish version of the Obstetric Quality of Recovery-10 questionnaire (ObsQoR-10-T), measured by a blinded assessor. Scores range from 0 to 100, with higher scores indicating better recovery.

SECONDARY OUTCOMES:
Total Opioid Consumption in 24 Hours | 0-24 hours postoperatively
  Total intravenous morphine consumption (in milligrams) recorded from PCA device logs in the first 24 hours after surgery.
Numerical Rating Scale (NRS) Pain Scores | 0-24 hours postoperatively
  Pain intensity measured using a Numerical Rating Scale (0 = no pain, 10 = worst pain imaginable) at specified postoperative time points.
Time to First Breastfeeding | Assessed from end of surgery to first breastfeeding attempt, up to 24 hours
  Time interval in minutes from the completion of surgery to initiation of breastfeeding.
Time to First Mobilization | Assessed from the end of surgery to first mobilization attempt, up to 24 hours postoperatively
  Time interval in hours from completion of surgery to the first mobilization with assistance or independently.
Time to Hospital Discharge | Assessed from the end of surgery to official hospital discharge, up to 7 days postoperatively
  Time interval from the end of surgery until the patient is formally discharged from hospital care.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Gökhan Taflan, MD, Principal Investigator — Samsun Education and Research Hospital
Locations (1):
- Samsun University Training and Research Hospital, Samsun, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD), data dictionary, and statistical analysis code will be shared with qualified researchers upon reasonable request, after publication of the main results. Data will be available 12 months after study completion and for up to 5 years. Requests must be accompanied by a methodologically sound proposal and relevant ethics approval.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: IPD and supporting information will be available beginning 12 months after the study's completion date and remain available for 5 years.
Access Criteria: Qualified researchers affiliated with academic institutions or research organizations, who provide a methodologically sound proposal and relevant ethics approval, may request access. Requests will be reviewed by the principal investigator. Approved researchers will receive access to de-identified datasets and related documentation via secure institutional data sharing platforms.